CLINICAL TRIAL: NCT00184990
Title: Effect of Selective iNOS Inhibition During Human Endotoxemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PP01
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-04

CONDITIONS: Endotoxemia
Keywords: Endotoxemia; Aminoguanidine
MeSH Terms: conditions — Endotoxemia | interventions — pimagedine; Endotoxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Aminoguanidine
Drug: endotoxin

SUMMARY:
Sepsis or endotoxemia is manifested by hypotension, resistance to vasopressors, myocardial depression,and altered organ blood flow distribution. The mechanisms underlying the cardiovascular dysfunction during sepsis are complex; however, they are partially mediated by an uncontrolled production of NO by inducible NO synthase (iNOS).Control subjects received 2 ng/kg E. coli endotoxin, whereas the active intervention group received endotoxin in the presence of selective iNOS-inhibitor aminoguanidine. Hemodynamics, vascular responses to norepinephrine, acetylcholine and sodium nitroprusside, as well as circulating cytokines and other mediators of inflammation were measured. We tested the hypothesis that inhibition of NO-synthesis prevented the LPS-mediated insensitivity to noradrenalin and endothelial-dependent vasorelaxation. Furthermore, we tested whether NO participates in occurrence of the endotoxin tolerance in humans by using the iNOS inhibitor aminoguanidine on healthy volunteers with endotoxemia. At 0; 2 and 4 hours after the LPS challenge whole blood was stimulated with five TLR agonists in vitro and pro- and anti-inflammatory cytokines were measured.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* tendency towards fainting
* alcohol abuse
* nicotine abuse
* drugs abuse

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2005-01; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Hemodynamics | 24 hrs after LPS administration
Markers of Inflammation | 24 hrs after LPS administration
Cytokines | 24 hrs after LPS administration
Markers of Renal Injury | 24 hrs after LPS administration
Inducible NO synthase expression | 24 hrs after LPS administration
NO-metabolites | 24 hrs after LPS administration
Mediators of Vascular reactivity | 24 hrs after LPS administration
Sensitivity to norepinephrine | 24 hrs after LPS administration
Endothelial-dependent vasorelaxation | 24 hrs after LPS administration

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pickkers, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands